CLINICAL TRIAL: NCT03578471
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application
Brief Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application - 2018_16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_16
Record Dates: First submitted 2018-06-20; First posted 2018-07-06 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Hearing Loss; Normal Hearing
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hearing Aid without NR and BF (Active Comparator): Hearing Aid without Noise Reduction (NR) or beam forming (BF) enabled serves as reference condition.
  Interventions: Device: Hearing Aid without NR and BF
- Hearing Aid with NR (Experimental): Hearing Aid with Noise Reduction (NR) enabled.
  Interventions: Device: Hearing Aid with NR
- Hearing Aid with BF (Experimental): Hearing Aid with beam forming (BF) enabled.
  Interventions: Device: Hearing Aid with BF

INTERVENTIONS:
Device: Hearing Aid without NR and BF — Each participant will be fitted with the Noise Reduction (NR) and Beamforming (BF) disabled. Disabled means that no sound processing algorithm that removes noise from the speech signal is active.
  Arms: Hearing Aid without NR and BF
Device: Hearing Aid with NR — Each participant will be fitted with the Noise Reduction (NR)(Sound Changing) program on the same hearing aid. Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort. The Noise Reduction is working spatially independent.
  Arms: Hearing Aid with NR
Device: Hearing Aid with BF — Each participant will be fitted with a beam forming program on the same hearing aid. Beam forming (BF) principle is a sound processing algorithm to remove noise from certain directions to improve the speech intelligibility and comfort.
  Arms: Hearing Aid with BF

SUMMARY:
An EEG study using continuous speech stimuli to assess neural language processing in a hearing impaired population. Participants listen to short radio excerpts in different Signal to Noise Ratios (SNR) and answer comprehension questions as well as listening effort questions. We assess the effect of different algorithms on neural language processing as well as subjective listening effort. Each participant hears 12 randomized segments of speech (about 4min long each) with different settings on their hearing aid (reference condition, noise reduction algorithm, beam forming algorithm). This will be a controlled, single blinded and randomized active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarter based in Stäfa.

ELIGIBILITY:
Inclusion Criteria:

* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) data | 8 weeks
  Neural language processing will be assessed through the EEG data collected while the participant is listening to running speech (neurophysiological data). Analysis of the brainstem response, cortical entrainment, N400 and alpha power are planned. EEG data is measured in Volt (mV), and entrainment data is analysed through coherence (frequency-based measure of correlation between the acoustic and the neural signal). N400 and alpha power are measured on the variance of mV over time.

SECONDARY OUTCOMES:
Subjective Listening Effort rating | 8 weeks
  The subjective Listening Effort rating will be assessed through self-reported individual listening effort on a scale from "extreme effort" to "no effort".

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Raether, Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No